CLINICAL TRIAL: NCT04801693
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 1819479 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled Parallel Group Design) and Effect of Food on the Relative Bioavailability of BI 1819479 (Open-label, Randomised, Two-way Crossover Design)
Brief Title: A Study in Healthy Men to Test How Well Different Doses of BI 1819479 Are Tolerated and Taken up by the Body With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1462-0001; 2021-000208-39 (EudraCT Number)
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: single rising dose part is single-blind, randomized, placebo-controlled within parallel dose groups.
  food effect part is randomized, open-label, two-way, two-period, crossover design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BI 1819479 (Experimental): single rising doses (SRD) part
  Interventions: Drug: BI 1819479
- Placebo (Placebo Comparator): Single rising doses (SRD) part
  Interventions: Drug: Placebo
- BI 1819479 fed - fasted arm (Experimental): Food effect part
  Interventions: Drug: BI 1819479
- BI 1819479 fasted - fed arm (Experimental): Food effect part
  Interventions: Drug: BI 1819479

INTERVENTIONS:
Drug: BI 1819479 — BI 1819479
  Arms: BI 1819479; BI 1819479 fasted - fed arm; BI 1819479 fed - fasted arm
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main objectives of the single rising doses (SRD) trial part are to investigate safety, tolerability and pharmacokinetics (PK) of BI 1819479 in healthy male subjects following administration of single rising doses.

The main objective of the food effect part is to investigate the influence of food on the relative bioavailability of BI 1819479.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
2. Age of 18 to 50 years (inclusive)
3. BMI of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular, hepatic parameters (ALT/AST) or renal parameters (creatinine) exceeding the ULN after repeated measurements
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts -Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with drug-related adverse events | Up to Day 36
  Single rising doses (SRD) part
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to Day 31
  Food effect part
Maximum measured concentration of the analyte in plasma (Cmax) | Up to Day 31
  Food effect part

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | Up to Day 31
  SRD part
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to Day 31
  SRD part
Area under the concentration-time curve of the analyte over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to Day 31
  Food effect part

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com